CLINICAL TRIAL: NCT04461522
Title: Prospective Cohort Study on the Outcome of Treatment of Rotator Cuff Injury by Ultrasound-guided
Brief Title: Study on the Outcome of Treatment of Rotator Cuff Injury by Ultrasound-guided Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M20191203
Record Dates: First submitted 2020-05-07; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Rotator Cuff Injury
Keywords: rotator cuff injury; Ultrasound-guided drug injection
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group
  Interventions: Procedure: Ultrasound-guided drug injection
- Control group

INTERVENTIONS:
Procedure: Ultrasound-guided drug injection — The injection drugs were glucocorticoids and anesthetic drugs (1ml+2% lidocaine hydrochloride 0.5ml+0.9% sodium chloride 0.5ml), and the injection sites were subacromion deltoid bursa/coracoid bursa/biceps longhead tenosynosheath/glenohumeral joint bursa, etc.
  Groups: Exposed group

SUMMARY:
Rotator cuff injury is a common shoulder joint disease in clinic. If conservative treatment fails to improve pain symptoms and range of motion, the surgical indications are. Numerous studies have shown that the pain of rotator cuff injury usually comes not from the broken tendon, but from periarthritis tendonitis, bursitis or adhesive shoulder capsule, etc. Ultrasound-guided drug injection combined with conventional rehabilitation treatment can significantly improve the pain symptoms and increase joint mobility. This study intends to use prospective cohort study methods, exposed factors for ultrasound-guided injection drug treatment, establish a rotator cuff injury exposure group and the control group of shoulder joint dysfunction queue, whether of ultrasound guided drug injection therapy can increase the shoulder joint function analysis, and explore for the rotator cuff injury method provides the basis of the evidence-based conservative treatment. The establishment of a conservative treatment cohort for rotator cuff injury will also lay the foundation for the accurate rehabilitation treatment of rotator cuff injury.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint around shoulder joint discomfort or restricted movement
* Nuclear magnetic or ultrasound in the diagnosis of rotator cuff injury and not to consider surgery patients
* Assessed by the musculoskeletal ultrasound images, diagnosed with tendonitis around shoulder joint, slippery bursa phlogistic or adhesive shoulder level
* Section capsule, such as indications of patients treated with ultrasound guided by injection.

Exclusion Criteria:

* History of shoulder fractures, open trauma, or surgery combined with shoulder and hand syndrome, gout, autoimmune arthritis, infectious arthritis, and other factors resulting in shoulder pain or limited mobility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: He was admitted to the third hospital of Peking University due to the dysfunction of shoulder joint caused by rotator cuff injury
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder function | Beginning
  VAS
Shoulder function | 1 week
  VAS
Shoulder function | 1 month
  VAS
Shoulder function | 3months
  VAS
Shoulder function | 6 months
  VAS
Shoulder function | Beginning
  ROM
Shoulder function | 1 week
  ROM
Shoulder function | 1 month
  ROM
Shoulder function | 3months
  ROM
Shoulder function | 6 months
  ROM
Shoulder function | Beginning
  Constant Test
Shoulder function | 1 week
  Constant Test
Shoulder function | 1 month
  Constant Test
Shoulder function | 3months
  Constant Test
Shoulder function | 6 months
  Constant Test

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes